CLINICAL TRIAL: NCT03402204
Title: Efficacy of High-Dose and Low-Dose Simvastatin on Vascular Oxidative Stress and Neurological Outcomes in Patients With Acute Ischemic Stroke: A Randomized, Double-Blind, Parallel, Controlled Trial
Brief Title: Efficacy of High and Low-Dose Simvastatin on Vascular Oxidative Stress and Neurological Outcome in Patients With AIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Pannawat Chaiyawatthanananthn, Faculty of Medicine, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MTU-EC-IM-4-019/58
Record Dates: First submitted 2015-08-14; First posted 2018-01-18 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Ischemic Stroke
Keywords: Simvastatin; Plaque stability; Acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Simvastatin; ubenimex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin 10 mg (Experimental): Simvastatin 10 mg
  Interventions: Drug: Simvastatin 10 mg
- Simvastatin 40 mg (Experimental): Simvastatin 40 mg
  Interventions: Drug: Simvastatin 40 mg

INTERVENTIONS:
Drug: Simvastatin 10 mg — Simvastatin is a cholesterol-lowering medication that blocks the production of cholesterol (a type of fat) in the body.
  Simvastatin reduces low-density lipoprotein (LDL) cholesterol and total cholesterol in the blood. Lowering your cholesterol can help prevent heart disease and hardening of the arteries, conditions that can lead to heart attack, stroke, and vascular disease.
  Other Names: Bestatin
  Arms: Simvastatin 10 mg
Drug: Simvastatin 40 mg — Simvastatin is a cholesterol-lowering medication that blocks the production of cholesterol (a type of fat) in the body.
  Simvastatin reduces low-density lipoprotein (LDL) cholesterol and total cholesterol in the blood. Lowering your cholesterol can help prevent heart disease and hardening of the arteries, conditions that can lead to heart attack, stroke, and vascular disease.
  Other Names: Bestatin
  Arms: Simvastatin 40 mg

SUMMARY:
Patients with acute ischemic stroke will be divided into 2 groups by double-blind, randomized, and controlled trial. Personality and past history of the patients will be recorded after the patients signed inform consent. The patient will be collected blood among 10 cc. for measurement biomarker in serum that related plaque stability for baseline and obtained neurological examination for baseline.

The patients must be take pills for 180 days by randomized code number on pill box, and patients must be turn into the site for follow up visit at Day 90 and Day 180. All visits of the patients will be collected blood among 10 cc. for measurement biomarker in serum that related plaque stability and obtained neurological examination.

Next, the data will be separated with code number for divided group into 2 groups. Group 1 is simvastatin 10 mg per day treatment (n=36) and Group 2 is simvastatin 40 mg per day treatment. Finally, all data of each group will be calculated mean ± standard deviation, and compared by statistical analysis.

DETAILED DESCRIPTION:
Patients with acute ischemic stroke will be divided into 2 groups by double-blind, randomized, and controlled trial. Personality and past history of the patients will be recorded after the patients signed inform consent. The patient will be collected blood among 10 cc. for measurement biomarker in serum that related plaque stability i.e. sLOX-1 and NO levels for baseline and obtained neurological examination i.e. NIHSS, mRS and Barthel's index scale for baseline. The bloods will be centrifuged 4,000 rpm for 15 minutes at 4˚C. The supernatant will be collected for determine sLOX-1 and NO levels by ELIZA.

The patients must be take pills for 180 days by randomized code number on pill box, and patients must be turn into the site for follow up visit at Day 90 and Day 180. All visits of the patients will be collected blood among 10 cc. for measurement biomarker in serum that related plaque stability i.e. sLOX-1 and NO, and obtained neurological examination i.e. NIHSS, mRS and Barthel's index scale. The bloods were centrifuged 4,000 rpm for 15 minutes at 4˚C. The supernatant were collected for determine all biomarkers by ELIZA.

Next, the data will be separated with code number for divided group into 2 groups. Group 1 is simvastatin 10 mg per day treatment (n=36) and Group 2 is simvastatin 40 mg per day treatment (n=36) . Finally, all data of each group will be calculated mean ± standard deviation, and compared by statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute ischemic stroke has symptom onset less than 24 hours.
* Patient has 18 to 85 years old.
* Patient has been obtained describe the study and sign on informed consent.

Exclusion Criteria:

* Patient has indication for simvastatin or ya-hom-navakote.
* Patient has pre-stroke mRS score more than 1.
* Patient was enrolled in other study within 30 days ago.
* Researchers consider that could be harmed by the participants or have certain conditions that could affect the participation in research, such as last stage of cancer.
* According to medical research suggests that patients unable to cooperate in research or inappropriate in joint research with other causes.
* Conscious level has >2 scores on question 2 of NIHSS.
* Platelet counts have less than 100,000 cells per cubic milliliter.
* Hematocrit has less than 0.25
* Blood sugar (BS) has less than 60 mg/dl or more than 200 ml/dl or between 200 and 300 mg/dl and treated with diabetes drug until the BS levels have less than 200 mg/dl can include for the project before receive the researched drug.
* Patient with uncontrolled hypertension by measure systolic blood pressure (SBP) has more than 200 mmHg and/or diastolic blood pressure (DBP) has more than 110 mmHg before receive the researched drug or patient that receive aggressive treatment.
* Patient with others stroke or severe head injury within 6 weeks before enrolled to the project.
* Patient is received severe surgery within 14 days before enrolled to the project.
* Patient has seizure with acute ischemic stroke.
* Patient has acute myocardial infarction (AMI) or coronary heart disease (CHD) within 3 weeks before enrolled to the project.
* Patient who receives lower-lipid level drug i.e. Ezetrol, Fenofibrate, Gemfibrosil, and Niacin or statin drugs i.e. Atorvastatin and Pitavastatin.
* Patient has increasing liver enzyme level or liver abnormal disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2014-10-04 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
vascular oxidative stress by measuring Soluble lectin-like oxidized low density lipoprotein receptor-1 and Nitric oxide levels | 180 days
  Soluble lectin-like oxidized low density lipoprotein receptor-1 in microgram/milliliter and Nitric oxide in micromole/liter is biomarkers of vascular oxidative stress.

SECONDARY OUTCOMES:
neurological outcomes by measuring National Institutes of Health Stroke Scale (NIHSS) | 180 days
  NIHSS is a assessment of clinical neurology in stroke
neurological outcomes by modified Rankin's Scale (mRS) | 180 days
  mRS is a assessment of clinical neurology in stroke
neurological outcomes by measuring Barthel's index | 180 days
  Barthel's index is a assessment of clinical neurology in stroke

CONTACTS AND LOCATIONS:
Overall Officials: Sombat Muengtaweepongsa, M.D., Principal Investigator — Faculty of Medicine, Thammasat University

REFERENCES:
- [Derived] Uransilp N, Chaiyawatthanananthn P, Muengtaweepongsa S. Efficacy of High-Dose and Low-Dose Simvastatin on Vascular Oxidative Stress and Neurological Outcomes in Patient with Acute Ischemic Stroke: A Randomized, Double-Blind, Parallel, Controlled Trial. Neurol Res Int. 2018 Apr 18;2018:7268924. doi: 10.1155/2018/7268924. eCollection 2018. PMID 29850244